CLINICAL TRIAL: NCT04970498
Title: Application of MRI Quantitative Parameters in Identifying Myelosuppression Risk of Neoadjuvant Chemoradiotherapy for Rectal Cancer
Brief Title: Application of MRI in Identifying Myelosuppression Risk of Neoadjuvant Chemoradiotherapy for Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021111
Record Dates: First submitted 2021-06-30; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Rectal Cancer Stage II; Rectal Cancer Stage III
Keywords: Rectal Cancer; Myelosuppression; magnetic resonance imaging; IDEAL-IQ
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- acute myelosuppression group: WBC <4.0×10^9 14 days after radiotherapy
  Interventions: Diagnostic Test: MRI; Diagnostic Test: blood routine test
- chronic myelosuppression group: WBC <4.0×10^9 90 days after radiotherapy
  Interventions: Diagnostic Test: MRI; Diagnostic Test: blood routine test
- no myelosuppression group: WBC >4.0×10^9 during radiotherapy
  Interventions: Diagnostic Test: MRI; Diagnostic Test: blood routine test

INTERVENTIONS:
Diagnostic Test: MRI — MRI including T1WI, DWI sequence and IDEAL-IQ sequence before radiotherapy, 1-2 weeks after radiotherapy and 90 days after radiotherapy were performed
Diagnostic Test: blood routine test — The blood routine was collected before radiotherapy, 1 week, 2 weeks and 90 days after radiotherapy.

SUMMARY:
Rectal cancer patients who received neoadjuvant chemoradiotherapy in Peking University Third Hospital in 2021 are divided into acute myelosuppression group, chronic myelosuppression group and normal group. The differences of magnetic resonance parameters between the groups were compared. The risk identification model of acute and chronic myelosuppression after neoadjuvant chemoradiotherapy was established by clinical risk factors and quantitative parameters of magnetic resonance imaging, and the prediction efficiency of the model was evaluated.

DETAILED DESCRIPTION:
The patients with locally advanced rectal cancer diagnosed in Peking University Third Hospital and undergoing neoadjuvant chemoradiotherapy were collected. The basic information of patients (including age, sex, BMI, TNM stage of rectal cancer (T2, T3 stage)) was collected. The blood routine was collected before radiotherapy, 1 week, 2 weeks and 90 days after radiotherapy. MRI including T1WI, DWI sequence and IDEAL-IQ sequence before radiotherapy, 1-2 weeks after radiotherapy and 90 days after radiotherapy were performed, and the corresponding parameters were obtained. The white blood cell values and quantitative parameters of magnetic resonance (including T1WI, DWI signal intensity (b = 1000) and proton density fat fraction (PDFF) of sacrilium and proximal femur were collected. Patients were divided into acute myelosuppression group and non-acute myelosuppression group according to blood routine results 14 days after radiotherapy, and chronic myelosuppression group and non-chronic myelosuppression group according to blood routine results 90 days after radiotherapy. The magnetic resonance parameters difference between 1-2 weeks after radiotherapy and before radiotherapy, and the magnetic resonance parameters difference between 90 days after radiotherapy and before radiotherapy were calculated. By comparing the differences of clinical risk factors and quantitative parameters of MRI between the two groups, the meaningful variables were screened out, and the risk identification model of acute and chronic myelosuppression was established.

ELIGIBILITY:
Inclusion Criteria:

* From February 2021 to August 2022, patients with locally advanced rectal cancer were treated with neoadjuvant chemoradiotherapy in the Third Hospital of Peking University.
* There were blood routine before radiotherapy, 1 week, 2 weeks and 90 days after radiotherapy, and MRI examination including routine MRI sequence and IDEAL-IQ sequence before radiotherapy, 1-2 weeks and 90 days after radiotherapy.
* Each patient used the same chemotherapy regimen.

Exclusion Criteria:

* Patients with metabolic bone diseases such as hyperparathyroidism and Cushing's syndrome.
* Patients with history of pelvic radiotherapy or systemic chemotherapy.
* Patients with leukocytes below 4.0×10^9/L or long-term severe anemia before radiotherapy.
* Patients with tumor bone metastases; patients with pelvic trauma, fracture, and infectious diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From February 2021 to August 2022, patients with locally advanced rectal cancer were treated with neoadjuvant chemoradiotherapy in the Third Hospital of Peking University
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes of IDEAL-IQ sequence of MRI | 1-2 weeks after radiotherapy
  The differences of PDFF(%) between the acute myelosuppression group and no suppression group
Changes of T1WI sequence of MRI | 1-2 weeks after radiotherapy
  The differences of T1WI signal intensity（IU） between the acute myelosuppression group and no suppression group
Changes of DWI sequence of MRI | 1-2 weeks after radiotherapy
  The differences of DWI signal intensity（IU）between the acute myelosuppression group and no suppression group
Changes of ADC map of MRI | 1-2 weeks after radiotherapy
  The differences of ADC value（mm^2/s) between the acute myelosuppression group and no suppression group
Changes of IDEAL-IQ sequence of MRI | 90 days after radiotherapy
  The differences of PDFF(%) between the chronic myelosuppression group and no suppression group
Changes of T1WI sequence of MRI | 90 days after radiotherapy
  The differences T1WI signal intensity（IU）between the chronic myelosuppression group and no suppression group
Changes of DWI sequence of MRI | 90 days after radiotherapy
  The differences of DWI signal intensity（IU）between the chronic myelosuppression group and no suppression group
Changes of ADC map of MRI | 90 days after radiotherapy
  The differences of ADC value（mm^2/s) between the chronic myelosuppression group and no suppression group

CONTACTS AND LOCATIONS:
Overall Officials: Ning Lang, Professor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No